CLINICAL TRIAL: NCT03804593
Title: HCCBloodTest for Detection of Hepatocellular Carcinoma (HCC): Marker Performance Validation and Technical Development Study
Brief Title: HCCBloodTest for Detection of Hepatocellular Carcinoma (HCC)
Status: Completed | Type: Observational
Sponsor: Epigenomics, Inc (Industry)
Collaborators: Innovis LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: Epigenomics 2018-HCC-A
Record Dates: First submitted 2019-01-11; First posted 2019-01-15 (Actual); Last update posted 2020-01-30 (Actual); Status verified 2020-01

CONDITIONS: Cirrhosis, Liver; Hepatic Cirrhosis; Hepatocellular Carcinoma; Liver Cancer
MeSH Terms: conditions — Liver Cirrhosis; Carcinoma, Hepatocellular; Liver Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — De-identified, clinically characterized plasma specimens for a bio-repository will be retained for up to twenty (20) years for future HCC-related test development.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: Diagnosis of cirrhosis and no HCC confirmed by medical imaging including MRI or CT performed within 6 months of study enrollment. If lesions are present, a Liver Imaging Reporting and Data System (LI-RADS) score of LR-1 or LR-2.
- Group 2: Diagnosis of HCC confirmed by medical imaging (MRI or CT performed within 6 months of study enrollment with LI-RADS score of LR-5) and/or biopsy with histopathology.

SUMMARY:
This is a multi-center study to prospectively gather clinically-characterized plasma samples to determine the diagnostic performance characteristics (sensitivity and specificity) of the HCCBloodTest among patients with cirrhosis with and without HCC

DETAILED DESCRIPTION:
Patients with clinically-diagnosed cirrhosis without HCC (Group 1) and patients with early-stage HCC (Group 2) will be invited to participate in this study consisting of one visit for all subjects. At Visit 1, Day 0, after subjects have provided informed consent and HIPAA consent, demographics (age, gender, ethnicity), etiology of liver disease and medical history as well as a list of current medications will be obtained; inclusion and exclusion criteria will be reviewed; and subjects will be registered into the study and will undergo a venipuncture to obtain four (4) lavender top K2 ethylenediaminetetraacetic acid (EDTA) 10 millilitre (mL) tubes of blood.

The HCCBloodTest will be performed on the blood samples collected from study subjects by the Sponsor at its laboratory in Berlin, Germany, to determine the performance characteristics of the HCCBloodTest in the study population.

The HCCBloodTest is an in-vitro polymerase chain reaction (PCR) assay for the qualitative detection of Septin 9 gene methylation (SEPT9) in DNA isolated from 3.5 mL of patient plasma. The SEPT9 gene is a key regulator of cell division and tumor suppressor and the hypermethylation of the assessed marker site is associated with liver carcinogenesis.

Results from the HCCBloodTest will be not be provided to the investigators or study subjects and, therefore, will be not be used in clinical decision-making or impact clinical care of the study participants in any manner.

ELIGIBILITY:
Inclusion Criteria:

* Men or women age 18 years or older;
* Able to read, understand and sign informed consent to participate in study;
* Willing and able to provide written informed consent;
* Willing and able to meet all study requirements and undergo venipuncture to provide blood samples;
* Child-Pugh Score of A or B.

Group 1:

• Diagnosis of cirrhosis and no HCC confirmed by abdominal contrast-enhanced MRI or CT study performed < 90 days prior to the date of consent or an MRI performed ≤ 45 days after Visit 1. If lesions are present, a LI-RADS score of LR-1 or LR-2.

Group 2:

• Diagnosis of HCC confirmed by abdominal contrast-enhanced MRI or CT study performed < 90 days prior to the date of consent or an MRI performed ≤ 45 days after Visit 1 with LI-RADS score of LR-5 and/or biopsy with histopathology.

Exclusion Criteria:

Both Groups:

* Child-Pugh Score of C;
* Subject has undergone a colonoscopy, endoscopy or other invasive diagnostic procedure (other than venipuncture) during the 10 days prior to providing a blood sample for this study;
* Pregnancy;
* Breastfeeding;
* Currently undergoing dialysis;
* Currently receiving investigational treatments of any type;
* History of receiving any drug therapy, surgery or liver transplant for the treatment of HCC;
* Diagnosis of any non-HCC cancer (other than non-melanoma skin cancer) within past 5 years and/or currently undergoing treatment for any cancer;
* Any clinical condition, diagnosis, or social circumstance that, in the opinion of the Investigator, would be mean participation in the study would be contraindicated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible subjects will be men and women age 18 years or older. Study will enroll sufficient subjects to yield a minimum of 100 evaluable subjects in Group 1, a minimum of 100 evaluable subjects with de novo HCC and cirrhosis in Group 2 and up to 20 subjects with de novo HCC without cirrhosis in Group 2 - a total of up to 220 evaluable study subjects who meet all inclusion and exclusion criteria for these two groups.
Sampling Method: Non-Probability Sample
Enrollment: 175 (Actual)
Dates: Start 2018-12-17 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2019-10-31 (Actual)

PRIMARY OUTCOMES:
Rate of SEPT9 gene promoter methylation positivity in patients with cirrhosis, based on the HCCBloodTest. | 45 days
  The HCCBloodTest is an in-vitro PCR based assay for the qualitative detection of the methylation status of a SEPT9 gene promoter DNA sequence. Plasma will be prepared from blood samples collected from study subjects and will be tested by the Sponsor with HCCBloodTest at its laboratory in Berlin, Germany. Positivity based on PCR results will be reported for study subjects. Test performance characteristics including sensitivity and specificity will be reported for the study population.

CONTACTS AND LOCATIONS:
Overall Officials: Theo DeVos, Study Director — Epigenomics, Inc; Nick Potter, Study Director — Epigenomics, Inc
Locations (2):
- United States (2):
  - USC Keck Medical Center, Los Angeles, California
  - California Liver Research Institute, Pasadena, California

REFERENCES:
- [Derived] Lewin J, Kottwitz D, Aoyama J, deVos T, Garces J, Hasinger O, Kasielke S, Knaust F, Rathi P, Rausch S, Weiss G, Zipprich A, Mena E, Fong TL. Plasma cell free DNA methylation markers for hepatocellular carcinoma surveillance in patients with cirrhosis: a case control study. BMC Gastroenterol. 2021 Mar 25;21(1):136. doi: 10.1186/s12876-021-01714-8. PMID 33765926